CLINICAL TRIAL: NCT02067897
Title: Nonrandomized Assessment of Ingrown ToenaiLs Treated by Excision of Skinfold Rather Than Toenail (NAILTEST): a Study of the Vandenbos Procedure in Children and Adolescents
Brief Title: Nonrandomized Assessment of Ingrown ToenaiLs Treated by Excision of Skinfold Rather Than Toenail
Acronym: NAILTEST
Status: Unknown | Type: Observational
Last Known Status: Enrolling by invitation
Sponsor: Michael Livingston (Other)
Collaborators: The Physicians' Services Incorporated Foundation (Other)
Responsible Party: Sponsor-Investigator, Michael Livingston, Resident, Division of General Surgery, Western University, Canada
Organization: Western University, Canada (Other)
Other Study IDs: 104906
Record Dates: First submitted 2014-02-12; First posted 2014-02-20 (Estimated); Last update posted 2014-11-13 (Estimated); Status verified 2014-11

CONDITIONS: Nails, Ingrown
Keywords: Nails, Ingrown; Children; Ambulatory Surgical Procedures
MeSH Terms: conditions — Nails, Ingrown

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Vandenbos procedure (skinfold excision): Participants in this cohort will undergo with Vandenbos procedure (skinfold excision) for one or more ingrown toenails. This surgery will be formed as an day procedure under general anesthetic.

SUMMARY:
Ingrown toenails occur when the nail grows into the surrounding skin, resulting in pain and infection. The most common procedure to treat this problem is a wedge excision (removal of part of the toenail) and matricectomy (destruction of part of the nailbed with chemicals or surgical instruments). This study will evaluate the effectiveness of an alternative technique called the Vandenbos procedure (where the skin is removed and the toenail is left intact). This procedure is currently being used by some of the pediatric surgeons at our hospital and we want to evaluate our results up to 6 months after surgery. We believe that the true recurrence rate will be greater than 0% but that recovery time and morbidity will be acceptable to most patients.

DETAILED DESCRIPTION:
Ingrown toenails are common among adolescents and young adults with the big toe being the most commonly affected. The exact incidence is unknown. An ingrown toenail occurs when the nail traumatizes the surrounding skin, resulting in swelling, infection, and the generation of granulation tissue. This cycle causes the nail to embed itself even further into the surrounding tissues, leading to additional swelling and infection.

Many treatments have been proposed for this condition. Non-surgical options include soaking, wearing loose shoes, antibiotics, and specialized braces. While these treatments often provide short-term symptomatic relief, many people with ingrown toenails eventually need surgery. The most common surgical treatment is a wedge excision (removal of the ingrown part of the nail). Most clinicians perform a partial matricectomy at the same time (destruction of part of the underlying nailbed with chemicals or surgical instruments). This prevents recurrence (where the toenail becomes ingrown again). The rate of recurrence with the wedge excision and matricectomy is reported to be 12-50%.

An alternative surgical technique is the Vandenbos procedure, where the skinfold is excised and allowed to heal by secondary intention over a period of approximately 6 weeks. This approach theoretically involves more pain, a higher risk of post-operative bleeding (because it is initially an open wound), and a longer recovery time. Proponents of this technique argue that these short-term morbidities are justified given the low rate of recurrence and excellent long-term results.

The original case series published by Vandenbos in 1959 found a recurrence rate of 0%. Two recent case series published by doctors from Ontario reported the same finding, but it was unclear how many patients in their series were lost to follow-up. Other studies have reported positive results but with a recurrence rate of 7-20%. Thus, the true effectiveness of this procedure remains unclear. Furthermore, there is no high quality evidence to support one technique over the other. Even a recent Cochrane review of 24 randomized controlled trials could not reach any definitive conclusions as to which procedure (among other surgical options) is the most effective. Previous trials show significant heterogeneity and none have assessed the Vandenbos procedure specifically. As a result, many clinicians continue to use the wedge excision and matricectomy.

ELIGIBILITY:
Inclusion Criteria:

* 10 to 18 years old
* Undergoing Vandenbos procedure for one or more ingrown toenails
* Willing to complete assessments

Exclusion Criteria:

* Inability to understand English
* Severe medical co-morbidities

Ages: 10 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: The study population include children and adolescents aged 10 to 18 years with one or more ingrown toenails. They may have undergone previous surgical and/or non-surgical treatment for this condition.
Sampling Method: Non-Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2014-04; Primary Completion 2016-04 (Estimated); Study Completion 2016-04 (Estimated)

PRIMARY OUTCOMES:
Recurrence | Up to 6 months after surgery
  Clinical signs of recurrence will be assessed 1 month, 2 months, and 6 months after surgery.

SECONDARY OUTCOMES:
Pain, functional status, and quality of life | Baseline, 1 month, 2 months, 6 months after surgery
  Pain, functional status, and quality of life will be measured with the 5-item EuroQol-5D-5L.
Patient satisfaction | 6 months after surgery
  Patient satisfaction with the Vandenbos procedure will be measured with the 8-item Surgical Satisfaction Questionnaire (SSQ).
Recovery time | 1 month, 2 months, 6 months after surgery
  Recovery time will be calculated in days off before returning to work, school, and normal footwear.

CONTACTS AND LOCATIONS:
Overall Officials: Sarah A Jones, MD, PhD, FRCSC, Principal Investigator — Division of Pediatric Surgery
Locations (1):
- Children's Hospital of Western Ontario, London Health Sciences Centre, London, Ontario, Canada

REFERENCES:
- [Background] Yang G, Yanchar NL, Lo AY, Jones SA. Treatment of ingrown toenails in the pediatric population. J Pediatr Surg. 2008 May;43(5):931-5. doi: 10.1016/j.jpedsurg.2007.12.042. PMID 18485969
- [Background] Heidelbaugh JJ, Lee H. Management of the ingrown toenail. Am Fam Physician. 2009 Feb 15;79(4):303-8. PMID 19235497
- [Background] Eekhof JA, Van Wijk B, Knuistingh Neven A, van der Wouden JC. Interventions for ingrowing toenails. Cochrane Database Syst Rev. 2012 Apr 18;2012(4):CD001541. doi: 10.1002/14651858.CD001541.pub3. PMID 22513901
- [Background] Vandenbos KQ, Bowers WF. Ingrown toenail: a result of weight bearing on soft tissue. U S Arm Forces Med J 1959;10:1168-73.
- [Background] Chapeskie H, Kovac JR. Case Series: Soft-tissue nail-fold excision: a definitive treatment for ingrown toenails. Can J Surg. 2010 Aug;53(4):282-6. PMID 20646404
- [Background] Haricharan RN, Masquijo J, Bettolli M. Nail-fold excision for the treatment of ingrown toenail in children. J Pediatr. 2013 Feb;162(2):398-402. doi: 10.1016/j.jpeds.2012.07.056. Epub 2012 Sep 10. PMID 22974574
- [Background] Antrum RM. Radical excision of the nailfold for ingrowing toenail. J Bone Joint Surg Br. 1984 Jan;66(1):63-5. doi: 10.1302/0301-620X.66B1.6693479.
- [Background] Persichetti P, Simone P, Li Vecchi G, Di Lella F, Cagli B, Marangi GF. Wedge excision of the nail fold in the treatment of ingrown toenail. Ann Plast Surg. 2004 Jun;52(6):617-20. doi: 10.1097/01.sap.0000095436.08812.67. PMID 15167000
- [Background] Mitchell S, Jackson CR, Wilson-Storey D. Surgical treatment of ingrown toenails in children: what is best practice? Ann R Coll Surg Engl. 2011 Mar;93(2):99-102. doi: 10.1308/003588411X12851639107674. Epub 2010 Nov 12. PMID 21073822